CLINICAL TRIAL: NCT02095418
Title: Open Label, Multicenter Randomized Control Study to Investigate the Incidence of NODAT (New-Onset Diabetes After Transplantation), Safety and Efficacy of Corticosteroids Early Withdrawal in Liver Transplanted Recipients
Brief Title: Comparison of New-onset Diabetes After Transplantation Between Two Steroid Withdrawal Group With CellCept
Acronym: NODAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, JAE WON JOH, Coordinating Investigator, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML28170
Record Dates: First submitted 2014-03-14; First posted 2014-03-24 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Diabetes
Keywords: New-onset diabetes after transplantation (NODAT); Liver transplantation
MeSH Terms: conditions — Diabetes Mellitus | interventions — Mycophenolic Acid; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mycophenolate mofetil, Corticosteroids (Experimental): * Mycophenolate mofetil: 500-1500mg/day, bid, PO
  * Corticosteroids: 500mg for the first dosage. It will be tapered at least 5mg for 14days and withdrawn
  Interventions: Drug: Corticosteroids, Mycophenolate mofetil
- Corticosteroids, Mycophenolate mofetil (Active Comparator): * Mycophenolate mofetil: 500-1000mg/day, bid, PO
  * Corticosteroids 500mg for the first dosage. It will be tapered at least 5mg for 3months(± 2 weeks) and withdrawn.
  Interventions: Drug: Mycophenolate mofetil, Corticosteroids

INTERVENTIONS:
Drug: Mycophenolate mofetil, Corticosteroids — tacrolimus (low dose, trough level of 5-12ng/ml)+Mycophenolate mofetil(500-1500mg/day*, bid)+ Basiliximab + corticosteroids 500mg to 5mg or above (2 weeks)
  Other Names: CellCept, Methylon
  Arms: Corticosteroids, Mycophenolate mofetil
Drug: Corticosteroids, Mycophenolate mofetil — tacrolimus (low dose, trough level of 5-12ng/ml)+Mycophenolate mofetil(500-1000mg/day*, bid)+ Basiliximab + corticosteroids 500mg to 5mg or above (3 month±2weeks)
  Other Names: Methylon, CellCept
  Arms: Mycophenolate mofetil, Corticosteroids

SUMMARY:
With improvements in patient and graft survival, increasing attention has been placed on complications that contribute to long-term patient morbidity and mortality. New-onset diabetes after transplantation (NODAT) is a common complication of solid-organ transplantation, and is a strong predictor of graft failure and cardiovascular mortality in the transplant population. Risk factors for NODAT in transplant recipients are similar to those in non-transplant patients, but transplant-specific risk factors such as hepatitis C (HCV) infection, corticosteroids and calcineurin inhibitors play a dominant role in NODAT pathogenesis. The predominant factor for causing NODAT by corticosteroids seems to be the aggravation of insulin resistance; however several studies have displayed deleterious effects on insulin secretion and β-cells. Thus, adjusting the immunosuppressant regimen to improve glucose tolerance must be measured and defined from long term perspective.

As recipients of organ transplants survive longer, the complications of NODAT have assumed greater importance; therefore, we designed a prospective study to compare the safety and efficacy of early versus late withdrawal of corticosteroids after liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* 1.Male or female patients between 20-70 years 2.De novo patients 3.Recipients from living or cadaveric donors 4.Single organ recipient (liver only) 5.White Blood Cell(WBC) ≥ 3,000uL 6.Women of childbearing potential had to have a negative serum or urine pregnancy test within 1 week prior to beginning study treatment. Effective contraception has to be used before beginning therapy, during therapy and for 6 weeks following discontinuation of therapy 7.Patients co-operative and able to complete all the assessment procedures. 8.Patients provided written informed consent

Exclusion Criteria:

1. Patients who receive immunosuppressive therapy (except steroid treatment) within the preceding 28 days.
2. Incompatible A,B, and O blood group system.
3. Active infection
4. Patients whose laboratory results reveal severe anaemia (as defined by a haemoglobin value < 9 g/dL for adults receiving erythropoietin, 6.5 g/dL for adults not receiving erythropoietin, leukopenia (as defined by a white blood cell [WBC] value of <1500/mm3) or thrombocytopenia (as defined by a platelet count of <30,000/mm3).
5. Mandatory intake of prohibited drugs or if it is probable that the patient would require treatment with such drugs after transplant
6. Patient is allergic or intolerant to excipients, steroids, Mycophenolate mofetil(MMF), tacrolimus or basiliximab.
7. Patients with any form of substance abuse, psychiatric disorder or condition, which, in the opinion of the investigator, may invalidate communication with the investigator or with study procedures.
8. The receipt of a new investigational drug within the previous 3 months
9. Pregnant or lactating females.
10. Women of child-bearing potential not willing to use a reliable form of contraception.
11. Previous organ transplantation
12. Patients who have diabetes mellitus prior to transplantation
13. Patients who have cancer other than liver cancer
14. Patients who have HGPRT(hypoxanthine quinine phosphoribosyl transferase) deficiency, Lesch-Nyhan syndrome, Kelly-Seegmiller syndrome

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2014-02; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate incidence of NODAT in patients of two arms | for 1 year
  NODAT will be defined as consecutively FPG ≥126mg/dl in two different days or PPG 2hr ≥200mg/dl Ref. Steroid Withdrawal in Adult Liver Transplantation: Occurrence at a Single Center. Transplantation Proceedings, 2010; 42: 4132-4136)
  1. Incidence of NODAT in ref. : (9.9%)
  2. 95% Confidence Interval(CI): (6%)
  Considering 10% drop-out rate, 76 patients will be enrolled in one arm. Totally, 152 will be enrolled.

SECONDARY OUTCOMES:
To evaluate incidence rate of first acute rejection | for 1 year
To evaluate time to first acute rejection | for 1 year
To evaluate proportion of patients experiencing treatment failure | for 1 year
To evaluate graft survival rates | for 1 year
To evaluate patient overall survial, OS | for 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jae Won Joh, M.D., Ph.D., Principal Investigator — Samsung Medical Center; Kwang-Woong Lee, M.D., Ph.D., Principal Investigator — Seoul National University Hospital; Seoung Hoon Kim, M.D., Ph.D., Principal Investigator — National Cancer Center; Hee-Jung Wang, M.D., Ph.D., Principal Investigator — Ajou University School of Medicine; Dongrak Choi, M.D., Ph.D., Principal Investigator — Daegu Catholic University Medical Center
Locations (5):
- South Korea (5):
  - Daegu Catholic University Medical Center, Daegu
  - Samsung Medical Center, Seoul
  - National Cancer Center, Seoul
  - Seoul National University, Seoul
  - Ajou University Hospital, Suwon